CLINICAL TRIAL: NCT06727981
Title: Prospective Cohort Study on the Efficacy, Adverse Effects, and Biomarkers of First-Line/Neoadjuvant Therapy With Immune Checkpoint Inhibitors Combined With Chemotherapy in Advanced Gastric Cancer
Brief Title: First-Line and Neoadjuvant Immunotherapy for Gastric Cancer
Status: Recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Lian Liu, MD, PHD, Professor, Chief Physician, Qilu Hospital of Shandong University
Other Study IDs: EABI-GC
Record Dates: First submitted 2024-09-27; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Advanced Gastric Cancer; Locally Advanced Gastric Carcinoma
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Collect the peripheral blood and feces of patients before and after treatment, and obtain pathological sections if possible.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ICI plus chemotherapy
  Interventions: Drug: ICI plus Chemothearpy
- Chemotherapy
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: ICI plus Chemothearpy — This intervention involves the administration of immune checkpoint inhibitors (ICIs) in combination with standard chemotherapy.
  Groups: ICI plus chemotherapy
Drug: Chemotherapy — This intervention involves the administration of standard chemotherapy alone.
  Groups: Chemotherapy

SUMMARY:
This prospective observational study aims to evaluate the efficacy and safety of immune checkpoint inhibitors as first-line and neoadjuvant therapy for advanced gastric cancer, while also investigating relevant biomarkers to better understand their role in immunotherapy outcomes

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years old or above
2. Patients with advanced gastric cancer or locally advanced gastric cancer
3. Have not received any previous anti-tumor therapy
4. Patients expected to receive immunotherapy for first-line or neoadjuvant therapy
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
6. Adequate organ function

Exclusion Criteria:

1. Patients with contraindications to immunotherapy
2. Have received anti-tumor treatments such as immunotherapy and chemotherapy
3. Have a history of active immune deficiency or autoimmune diseases, including HIV positive test, or have other acquired or congenital immune deficiency diseases, or have a history of organ transplantation or autoimmune diseases
4. Severe chronic or active infection requires systemic antibacterial, antifungal, or antiviral treatment, including tuberculosis infection. Have a history of active tuberculosis infection ≥ 1 year before recruitment should also be excluded, unless proved has been completed appropriate treatment
5. History of allogeneic stem cell transplantation or organ transplantation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pathologically defined, locally inoperable or advanced gastric cancer who have not received any previous anti-tumor therapy and are expected to receive immunotherapy.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-01-15 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 12 months after the last subject participating in
  The time from the starting date of study drug to death

SECONDARY OUTCOMES:
Disease Control Rate (DCR) as assessed by RECIST1.1 | 6 months after the last subject participating in
  The proportion of subjects with complete response (CR) and partial response (PR) and stable disease(SD)in total subjects.
Duration of response (DOR) as assessed by RECIST1.1 | 12 months after the last subject participating in
  The time from the date for first documented response of complete response (CR) or partial response (PR) to the date of first documented of disease progression or death, whichever occurs first.
Number of participants with treatment-related adverse events as assessed by CTCAE5.0 | 12 months after the last subject participating in
  Incidence and severity of adverse effects associated with the treatments, categorized by type and grade according to the Common Terminology Criteria for Adverse Events (CTCAE v5.0).
Progression-free survival (PFS) as assessed by RECIST1.1 | 12 months after the last subject participating in
  The time from the starting date of study drug to the date of first documentation of disease progression or death, whichever occurs first
Objective remission rate (ORR) as assessed by RECIST1.1 | 3 months after the last subject participating in
  The proportion of subjects with complete response (CR) and partial response (PR) in total subjects
Disease-free survival (DFS) as assessed by RECIST1.1 | 36 months after the last subject participating in
  The period from treatment until the occurrence of disease recurrence, progression, or death.
Major pathological response (MPR) | 3 months after the last subject participating in
  he percentage of residual viable tumor cells in the resected specimen that is ≤10% after neoadjuvant therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Lian Liu, MD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No